CLINICAL TRIAL: NCT06774807
Title: Antagonist of the Glucagon-like Peptide 2 (GLP-2) Receptor
Brief Title: Blocking of the Gut Hormone Receptor for Glucagon-like Peptide 2 (GLP-2) by the GLP-2 Receptor Antagonist GLP-2(3-33)
Acronym: GLP-2ant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-24000668
Record Dates: First submitted 2025-01-07; First posted 2025-01-14 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Glucagon-Like Peptide 2; GLP-2; GLP-2 (3-33); GLP-2 (1-33); Gastrointestinal Blood Flow; Superior Mesenteric Artery; Portal Vein
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled, single-blinded, crossover-study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saline injection + Saline infusion (SAL-SAL) (Placebo Comparator): Saline subcutaneous injection, Intravenous saline infusion (NaCl (9 mg/ml))
  Interventions: Other: Saline infusion; Other: Saline injection
- GLP-2 agonist injection + Saline infusion (AGO-SAL) (Active Comparator): Subcutaneous injection of GLP-2 (1-33) agonist, Intravenous infusion of saline (NaCl (9 mg/ml))
  Interventions: Other: Saline infusion; Other: Agonist injection
- GLP-2 agonist injection + GLP-2 1 nmol antagonist infusion (AGO-1ANT) (Experimental): Subcutaneous Injection of GLP-2 (1-33) agonist, Intravenous infusion of 1 nmol/kg/min GLP-2 (3-33) antagonist
  Interventions: Other: 1nmol antagonist infusion; Other: Agonist injection
- GLP-2 agonist injection + GLP-2 4 nmol antagonist infusion (AGO-4ANT) (Experimental): Subcutaneous Injection of GLP-2 (1-33) agonist, Intravenous infusion of 4 nmol/kg/min GLP-2 (3-33) antagonist
  Interventions: Other: 4 nmol antagonist infusion; Other: Agonist injection

INTERVENTIONS:
Other: Saline infusion — Saline/NaCl (9mg/ml) intravenous infusion
  Arms: GLP-2 agonist injection + Saline infusion (AGO-SAL); Saline injection + Saline infusion (SAL-SAL)
Other: Saline injection — Saline/NaCl (9mg/ml) subcutaneous injection
  Arms: Saline injection + Saline infusion (SAL-SAL)
Other: 1nmol antagonist infusion — GLP-2 (1-33)/GLP-2(3-33) 1 nmol/kg/min
  Arms: GLP-2 agonist injection + GLP-2 1 nmol antagonist infusion (AGO-1ANT)
Other: 4 nmol antagonist infusion — GLP-2 (1-33)/GLP-2 (3-33) 4 nmol/kg/min
  Arms: GLP-2 agonist injection + GLP-2 4 nmol antagonist infusion (AGO-4ANT)
Other: Agonist injection — GLP-2(1-33) subcutaneous injection
  Arms: GLP-2 agonist injection + GLP-2 1 nmol antagonist infusion (AGO-1ANT); GLP-2 agonist injection + GLP-2 4 nmol antagonist infusion (AGO-4ANT); GLP-2 agonist injection + Saline infusion (AGO-SAL)

SUMMARY:
This project will describe the role of physiological levels of GLP-2 in regulating the blood flow to the intestines and the effect of the antagonist GLP-2(3-33) in blocking these effects of GLP-2.

DETAILED DESCRIPTION:
Ten healthy participants will meet fasting and attend four randomized experimental days of MRI-scans of the abdomen. Each day will include subcutaneous injections of GLP-2 or saline and intravenous infusion of either the GLP-2 (3-33) antagonist or saline. The infusion start at timepoint -20, while the subcutaneous injection is given to timepoint 0 and the participant will lay in the scanner in one hour after injection. Eight MR-scans are done repeatedly to measure the blood flow in larger abdominal vessels and four blood samples are taken during the experimental day for analysis of GLP-2(1-33), GLP-2(3-33) and bone markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* BMI 19-28 kg/m2

Exclusion Criteria:

* Chronic illness that affects the cardiovascular system or gastrointestinal tract
* Treatment with medicine or supplements that cannot be paused for 12 hours
* Intake of above 14 alcoholic drinks per week or substance abuse
* Liver enzymes (ALAT) above 2 times normal values
* Decreased kidney function (eGFR below 90 or creatinine levels over reference value)
* Low blood percentage (hemoglobin below reference value)
* Any condition or disease that the persons responsible for the study find would interfere with the participation of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-07 (Actual)

PRIMARY OUTCOMES:
SMA blood flow | 85 minutes
  Blood flow in the superior mesenteric artery

SECONDARY OUTCOMES:
PVblood flow | 85 minutes
  Blood flow in the portal vein

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Will be shared upon request

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT06774807/Prot_SAP_000.pdf